CLINICAL TRIAL: NCT03746704
Title: A Phase 1, First-in-Human Study of ImmunoPET Imaging of PD-L1 in Tumors Using 89Zr-DFO-REGN3504, an Anti-PD-L1 Tracer for Positron Emission Tomography in Patients With Advanced PD-L1 Positive Malignancies
Brief Title: Study of ImmunoPet Imaging of PD-L1 in Tumors Using 89Zr-DFO-REGN3504 in Adult Participants With Advanced PD-L1 Positive Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: R3504-ONC-1701
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Advanced PD-L1 Positive Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr˗DFO˗REGN3504 (Experimental): Part A: Cohorts 1-3 Part B
  Interventions: Drug: 89Zr˗DFO˗REGN3504

INTERVENTIONS:
Drug: 89Zr˗DFO˗REGN3504 — 89Zr˗DFO˗REGN3504

SUMMARY:
The primary objective of the study is to determine the safety and tolerability of 89Zr-DFO-REGN3504.

The secondary objectives of the study are:

Study Part A only:

* To establish adequate mass dose and activity dose of 89Zr˗DFO˗REGN3504 and optimal post-infusion imaging time, as assessed by imaging and blood draw after tracer infusion

Study Part B only:

* To establish test/re-test reliability of positron emission tomography (PET) measures as assessed on 2 separate tracer infusions at adequate mass dose and optimal imaging time point as determined in Part A
* To characterize the pharmacokinetic (PK) profile of 89Zr˗DFO˗REGN3504 based on tracer plasma activity concentration

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with at least 1 radiologically measurable (by RECIST 1.1) lesion (Note: Lesions 10 mm in diameter or larger at the high end Program Dealth-Ligand 1 (PD-L1) expression are expected to be detectable by 89Zr-DFO-REGN3504 PET imaging).
* Availability of an archival, formalin-fixed, paraffin-embedded (FFPE) tumor tissue sample (blocks or slides) from a primary/metastatic/recurrent site, which has not been previously irradiated, with presence of any PD-L1 expression by Immunohistochemistry (IHC) in tumor or immune cells, performed by a Clinical Laboratory Improvement Amendments of 1988 (CLIA), a certified laboratory, using either freshly cut or archived FFPE slides. If the analysis will be done using archived FFPE slides, the slides must be <6 months old after being cut from the tissue block. The age of a tissue block is not limited. If the patient has a report of ≥1% PD-L1 expression, there is no need to repeat the assay; the report has no time limit.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 (Oken, 1982) and anticipated life expectancy of at least 3 months
* Adequate organ and bone marrow function

Key Exclusion Criteria:

* Participants receiving therapy with a monoclonal antibody against PD-L1 (eg. durvalumab, atezolizumab, avelumab) or have received treatment with anti-PD-L1 within 135 days prior to the 89Zr˗DFO˗REGN3504 infusion date
* For Part B only, participants in whom anti-PD-1 therapy was initiated 1 month or less, prior to the 89Zr˗DFO˗REGN3504 infusion date
* Active or untreated brain metastases or spinal cord compression. Participants are eligible if the central nervous system (CNS) metastases are adequately treated and participants' neurological symptoms have returned to baseline levels (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. Participants with brain metastases must be off doses of corticosteroid therapy that are considered by the investigator to be immunosuppressive
* Known history of human immunodeficiency virus or known acquired immunodeficiency syndrome indicating uncontrolled active infection. Participants on highly active antiretroviral therapy with undetectable RNA levels and CD4 counts above 350 are permitted
* Receipt of an investigational compound or device within 30 days of screening or within 5 half-lives of the investigational compound or therapy being studied (whichever is greater)
* Major surgery or significant traumatic injury within 4 weeks prior to first dose of 89Zr˗DFO˗REGN3504
* Known psychiatric or substance abuse disorder, including current use of any illicit drugs, that would interfere with the participant's participation in, or compliance with the requirements of, the study
* History of hypersensitivity response to any protein therapeutics (eg, recombinant proteins, vaccines, IV immune globulins, monoclonal antibodies, receptor traps). If a patient intends to receive a COVID-19 vaccine during Part A only, participation in the dose-escalation part of the study should be delayed at least 1 week after the final dose of COVID-19 vaccine before the start of study drug.
* Sexually active men and women of childbearing potential who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose.
* Part B only: Has been enrolled in Part A

Note: Other Protocol Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Baseline through 90 days after last dose of tracer infusion

SECONDARY OUTCOMES:
Standardized uptake value (SUV) of 89Zr˗DFO˗REGN3504 in the blood pool | Up to day 8
  Part A
Clinical dosimetry based on the equivalent dose of radiation | Up to day 8
  Part A
Clinical dosimetry based on the effective dose of radiation | Up to day 8
  Part A
SUVs across the tumor region of interest (ROIs) | Up to day 8
  Part A
Maximal SUVs (SUVmax) within tumor ROIs | Up to day 8
  Part A
Pharmacokinetics (PK) of 89Zr˗DFO˗REGN3504; plasma tracer activity concentration of area under the curve (AUC0-7) | Up to day 8
  Part A
Change in SUV of 89Zr˗DFO˗REGN3504 in the blood pool | Up to day 36 ± 14 days
  Part B
Change in SUVs across the tumor ROIs | Up to day 36 ± 14 days
  Part B
Change in SUVmax within the tumor ROIs | Up to day 36 ± 14 days
  Part B
Biodistribution of 89Zr˗DFO˗REGN3504 | Up to day 36 ± 14 days
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/